CLINICAL TRIAL: NCT00326209
Title: A Multicenter, Open-Label, Treatment Extension Trial to Evalaute the Long-Term Safety and Tolerability of Mesalamine Pellet Formulation
Brief Title: Long-Term Safety and Tolerability of Mesalamine Pellets in Participants With Ulcerative Colitis in Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPUC3005
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Ulcerative Colitis
Keywords: UC; Ulcerative colitis; Inflammatory bowel disease; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

ARMS (1):
- Encapsulated Mesalamine Granules (eMG) (Experimental): Participants will receive eMG 1.5 grams (4 capsules of eMG 0.375 grams each) QD orally in the morning for up to 24 months.
  Interventions: Drug: Encapsulated Mesalamine Granules (eMG)

INTERVENTIONS:
Drug: Encapsulated Mesalamine Granules (eMG) — eMG capsules will be administered per dose and schedule specified in the arm.
  Other Names: Mesalamine pellets

SUMMARY:
To evaluate the long-term safety and tolerability of encapsulated mesalamine Granules (eMG) (formerly referred to as Mesalamine Pellets [MP]) in participants with ulcerative colitis currently in remission.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, open-label, treatment extension study evaluating the long-term safety and tolerability of eMG given once daily (QD) in participants who successfully participated in a double-blind lead-in study (MPUC3003 [NCT00744016 ] or MPUC3004 [NCT00767728 ]) or new participants who are currently in remission from symptoms of ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB)/Ethics Committee (EC) approved informed consent is signed and dated prior to any study-related activities.
2. Participant has successfully participated in a previous MP clinical study per investigator's discretion with successful participation minimally defined as compliant with study-related procedures and study drug dosing schedule in the previous study and did not discontinue from the previous study due to study drug-related AE(s) or if new participants:

   a. Participant is a male or,

   If the participant is female, she is eligible to enter if she is of:

   Non-childbearing potential (that is; physiologically incapable of becoming pregnant, including any female who has undergone sterilization [hysterectomy or bilateral tubal ligation] or is post-menopausal. For purposes of this study, postmenopausal is defined as 1 year without menses); or childbearing potential, has a negative serum pregnancy test at screen and, if heterosexually active, agrees to one of the following:

   i) Double barrier method of contraception, specifically, use of a condom and spermicide, for 1 week prior to study drug administration, throughout the 6-month Treatment Phase, and the 2-week follow-up phase.

   ii) Oral contraceptives administered for at least 2 monthly cycles prior to study drug administration during all 6 months of study drug administration and administered for 1 monthly cycle following completion of the study.

   iii) An intrauterine device (IUD), inserted by a qualified clinician, with published data showing that the lowest expected failure rate is less than (<)1% per year (not all IUDs meet this criterion).

   iv) Medroxyprogesterone acetate (DEPO-PROVERA) administered for a minimum of 1 monthly cycle prior to the study drug administration, during all 6 months of study drug administration, and administered for 1 monthly cycle following study completion. Norelgestromin/ ethinyl estradiol transdermal system (Ortho Evra patch) administered for at least 2 monthly cycles prior to study drug administration and administered for 2 monthly cycles following study completion.

   v) Partner has undergone vasectomy and participant is in a monogamous relationship.

   The investigator is responsible for determining whether the participant has adequate birth control for study participation.

   b. Participant is greater than or equal to (≥) 18 years of age. c. Participant has historically confirmed diagnosis (physician letter for newly/recently diagnosed and by medical records for previously diagnosed participants) of mild to moderate UC in remission for greater than (>) 1 month and <12 months.

   d. Confirmed current remission defined as both: A screening rectal bleeding score of 0 as described in the Disease Activity Index (DAI) (Sutherland Index) where 0 = None A screening sigmoidoscopy score of 0 to 1 for mucosal appearance as described in the (Sutherland Index where 0 = intact mucosa with preserved or distorted vessels and 1 = Erythema, decreased vascular pattern, granularity, no mucosal hemorrhage.
3. Participant and investigator consider there is the potential for benefit to the participant with MP treatment.
4. Participant is capable and willing to comply with all study procedures.

Exclusion Criteria:

1. Participant has any condition or circumstance that would, in the opinion of the investigator, prevent completion of the study or interfere with analysis of study results, including history of noncompliance with treatments or visits.

   If a new participant, the following additional exclusion criteria will apply:
2. Participant has a history of allergy or intolerance to aspirin, mesalamine or other salicylates.
3. Participant has an abnormal clinical lab result which in the opinion of the investigator is significant enough to prevent participant's enrollment in the study.
4. Participant or participant's parents are known to have phenylketonuria.
5. Participant has participated in an investigational drug or device study within the 30 days prior to study screening.
6. Participant shows evidence of current excessive alcohol consumption or drug dependence.
7. Participant has uncontrolled, clinically significant renal disease manifested by 1.5 * ULN of serum creatinine or blood urea nitrogen (BUN) levels.
8. Participant has calculated creatinine clearance level of <60 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2005-12-22 (Actual); Primary Completion 2008-05-05 (Actual); Study Completion 2008-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (61):
- United States (61):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - First Care Family Doctors South, Fayetteville, Arkansas
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - AGMG Clinical Research, Anaheim, California
  - Lovelace Scientific Resources, Beverly Hills, California
  - Digestive Liver Disease Specialists, Medical Group, Garden Grove, California
  - Long Beach VA Medical Center, Long Beach, California
  - Community Clinical Trials, Orange, California
  - Rider Research Group, San Francisco, California
  - John Jolley, M.D., San Rafael, California
  - Lovelace Scientific Resources, Santa Ana, California
  - Santa Barbara Clinical Research, Santa Barbara, California
  - Professionals for Clinical Research, Littleton, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Clinical Research of Tampa Bay, Inc., Brooksville, Florida
  - Medical Research Unlimited, Hialeah, Florida
  - Southern Clinical Research Consultants, Hollywood, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Venture Research Institute, LLC, North Miami Beach, Florida
  - Penninsula Research, Inc., Ormond Beach, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Advent Clinical Research, Sarasota, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Consultative Gastroenterology, Atlanta, Georgia
  - Digestive Care Associates, Austell, Georgia
  - Center for Gastroenterology, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Northwest Gastroenterologists S.C., Arlington Heights, Illinois
  - Covenant Clinic, Waterloo, Iowa
  - Cotton-O'Neil Digestive Health Center, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Sinai Medical Office Building, Baltimore, Maryland
  - Philip J. Beam Medical Center, Hollywood, Maryland
  - Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive & Liver Diseases, Mexico, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Shore Health Group, Ocean City, New Jersey
  - Simon Lichtiger, M.D., New York, New York
  - VA Medical Center, Northport, Northport, New York
  - VA Medical Center, Syracuse, New York
  - Upstate Gastroenterology Associates, PC, Troy, New York
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Bethany Medical Center, High Point, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - Consultants for Clinical Research, Inc., Cincinnati, Ohio
  - Avamar Center for Endoscopy, Warren, Ohio
  - Oklahoma Gastroenterology Associates, LLC, Tulsa, Oklahoma
  - Charleston Gastroenterology Specialists, LLC, Charleston, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Medical Research Institute, Nashville, Tennessee
  - NationsMed Clinical Research, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Houston Digestive Disease Clinic, Houston, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - New River Research Institute, Christiansburg, Virginia
  - Seattle Gastroenterology Associates, Seattle, Washington
  - Eastern Washington Clinical Research Center, Spokane, Washington
  - Spokane Digestive Disease Center, Spokane, Washington
  - Digestive Disease Research Center, Tacoma, Washington
  - Center for Advanced Research, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Lichtenstein GR, Gordon GL, Zakko S, Murthy U, Sedghi S, Pruitt R, Barrett AC, Bortey E, Paterson C, Forbes WP. Long-Term Benefit of Mesalamine Granules for Patients Who Achieved Corticosteroid-Induced Ulcerative Colitis Remission. Dig Dis Sci. 2016 Jan;61(1):221-9. doi: 10.1007/s10620-015-3866-7. Epub 2015 Nov 12. PMID 26563167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled participants were rolled over from a double-blind lead-in study (MPUC3003 [NCT00744016 ] or MPUC3004 [NCT00767728 ]), or were new participants with demonstrated remission of ulcerative colitis (UC) were enrolled in this study.
Pre-assignment Details: A total of 393 participants were enrolled into the study. Of the participants included in the study, 280 participants were rolled over from a lead-in study (MPUC3003 or MPUC3004) and 113 were new participants.
Groups:
- Encapsulated Mesalamine Granules (eMG): Participants received eMG 1.5 grams (4 capsules of eMG 0.375 grams each) once daily (QD) orally in the morning for up to 24 months.
Period: Overall Study
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Started | 393
Safety Population (Received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.) | 388
Completed | 111
Not Completed | 282
Not completed — Adverse Event | 28
Not completed — Withdrawal by Subject | 22
Not completed — Lack of Efficacy | 31
Not completed — Lost to Follow-up | 18
Not completed — Participant non-compliant | 6
Not completed — Sponsor closed study | 173
Not completed — Prohibited medication use | 1
Not completed — Violation of entry criteria | 1
Not completed — Withdrawn in error | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.
Groups:
- Encapsulated Mesalamine Granules (eMG): Participants received eMG 1.5 grams (4 capsules of eMG 0.375 grams each) QD orally in the morning for up to 24 months.
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Number analyzed (Participants) | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.6)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 342
  ≥65 years | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203
  Male | 185
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 226
  Russia | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A TEAE was defined as any event with a start date occurring on or after treatment Day 1 or, if pre-existing, worsening after treatment Day 1. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 1) up to follow-up (24.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Number analyzed (Participants) | 388
Participants | 280

2. Primary Outcome: Number of Participants Who Prematurely Discontinued Treatment
Description: Number of participants who prematurely discontinued treatment due to any reason were reported.
Time Frame: Baseline up to Month 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Number analyzed (Participants) | 388
Participants | 282

3. Primary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Hematology and Blood Chemistry Abnormalities
Description: Criteria for potentially clinically significant abnormal hematology and blood chemistry values included: hemoglobin (grams/deciliter [g/dL]): <10 and ≥3 decrease, or >20; hematocrit (%): <30 and ≥10 decrease, or >60; platelets (*10^9 cells/liter): <100 or >700 (normal: 150-400); white blood cells (*10^9 cells/liter): <2.3 or >16.2 (normal: 3.5-11.1); alanine aminotransferase (units/liter [U/L]): ≥3 * upper limit of normal (ULN) (normal range 0-47 U/L); aspartate aminotransferase (U/L): ≥3 * ULN (normal range 0-37 U/L); total bilirubin (micromoles/liter [µmol/L]): >2 times; and calcium creatinine clearance (milliliters/minute [mL/min]): ≤50.
Time Frame: Baseline up to follow-up (24.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Number analyzed (Participants) | 388
Participants
  Hemoglobin (g/dL) | 8
  Hematocrit (%) | 7
  Platelets (*10^9 cells/L) | 5
  White blood cells (*10^9 cells/L) | 13
  Alanine aminotransferase (U/L) | 3
  Aspartate aminotransferase (U/L) | 3
  Total bilirubin (µmol/L) | 6
  Calcium creatinine clearance (mL/min) | 2

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included systolic and diastolic blood pressure, pulse rate, body temperature, or body weight.
Time Frame: Baseline, up to follow-up visit (Month 24.5)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Number analyzed (Participants) | 388
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up (24.5 months)
Description: Safety population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment.
Arm/Group | Encapsulated Mesalamine Granules (eMG)
Serious Adverse Events (participants affected / at risk) | 28/388
Other Adverse Events (participants affected / at risk) | 280/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Encapsulated Mesalamine Granules (eMG) (N=388)
Periproctitis (Gastrointestinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Colitis ulcerative (Gastrointestinal disorders) | 6
Diverticular perforation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Abscess limb (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/203 — This is a gender-specific AE. Only female participants were at risk.
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/203 — This is a gender-specific AE. Only female participants were at risk.
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1/203 — This is a gender-specific AE. Only female participants were at risk.
Uterine perforation (Reproductive system and breast disorders) | 1/203 — This is a gender-specific AE. Only female participants were at risk.
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Encapsulated Mesalamine Granules (eMG) (N=388)
Diarrhea (Gastrointestinal disorders) | 42
Abdominal Pain (Gastrointestinal disorders) | 31
Colitis ulcerative (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 16
Haemorrhoids (General disorders) | 16
Vomiting (Gastrointestinal disorders) | 16
Abdominal pain upper (Gastrointestinal disorders) | 14
Abdominal distension (Gastrointestinal disorders) | 13
Haematochezia (Gastrointestinal disorders) | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12
Nasopharyngitis (Infections and infestations) | 54
Sinusitis (Infections and infestations) | 28
Upper respiratory tract infection (Infections and infestations) | 26
Gastroenteritis viral (Infections and infestations) | 19
Influenza (Infections and infestations) | 19
Respiratory tract infection viral (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 17
Bronchitis (Infections and infestations) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 26
Headache (Nervous system disorders) | 45
Insomnia (Psychiatric disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.